CLINICAL TRIAL: NCT06017882
Title: Combined Effects of Acute Sleep Restriction and Moderate Acceleration (+Gz) on Physiological and Behavioral Responses to High Mental Workload
Acronym: CogPhyAero
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: 2023PBMD06; 2023-A01101-44 (Other: IDRCB)
Record Dates: First submitted 2023-08-11; First posted 2023-08-30 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Sleep Deprivation
Keywords: acceleration; mental workload; aerospace medicine
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group A : Usual sleep *2 ; Deprivation *2: V1->V3 id. V4 : Usual sleep and test series (easy; difficult; difficult) V5 : Usual sleep and test series (difficult; easy; easy) V6 : Sleep deprivation and test series (easy; easy; difficult) V7 : Sleep deprivation and test series (difficult; difficult; easy)
  Interventions: Other: Partial sleep deprivation
- Group B : Usual sleep ; Deprivation; Deprivation ; Usual sleep: V1->V3 id. V4 : Usual sleep and test series ( difficult; difficult ; easy) V5 : Sleep deprivation and test series (easy; difficult; difficult) V6 : Sleep deprivation and test series (difficult; easy; easy) V7 : Usual sleep and test series (easy ; easy ; difficult)
  Interventions: Other: Partial sleep deprivation
- Group C : Deprivation; Usual sleep ; Deprivation ; Usual sleep: V1->V3 id. V4 : Sleep deprivation and test series (easy; easy; difficult) V5 : Usual sleep and test series (difficult; difficult; easy) V6 : Sleep deprivation and test series (easy; difficult; difficult) V7 : Usual and test series (difficult; easy; easy)
  Interventions: Other: Partial sleep deprivation
- Group D : Deprivation ; Deprivation ; Usual sleep ; Usual sleep: V1->V3 id. V4 : Sleep deprivation and test series (difficult; easy; easy) V5 : Sleep deprivation and test series (easy; difficult; easy) V6 : Usual sleep and test series ( difficult; easy ; easy) V7 : Usual sleep and test series (easy ; difficult; difficult)
  Interventions: Other: Partial sleep deprivation

INTERVENTIONS:
Other: Partial sleep deprivation

SUMMARY:
Fighter pilots have to perform tasks requiring high mental workload during moderate-intensity acceleration phases (2 to 3G) that can last several minutes. When these accelerations are performed in the body axis (+Gz), they induce a redistribution of blood flow in the lower limbs associated with a decrease in cerebral blood flow, partially compensated by activation of the sympathetic nervous system (baroreflex).

The main hypothesis is that the effects of these prolonged accelerations, even of moderate intensity (<+4Gz), could impair pilots' ability to perform complex cognitive tasks, with potential consequences for flight safety and mission conduct.

Moreover, flight missions are often performed after sleep debt, which is known to induce cardiovascular responses, sympathetic nervous system activation and impaired mental performance.

The secondary hypothesis is that sleep debt (3h of time spent in bed) may increase the impairment of cognitive performance during prolonged acceleration.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject (male or female);
* Tobacco consumption < 5 cigarettes per day or nicotine-free vapour;
* Regular physical activity (between 1 and 8 hours per week);
* Affiliated or entitled to a social security scheme;
* Having given their consent.

Exclusion Criteria:

* Presenting an active medical pathology or a history <6 months (cardiological, renal, hepatic, cutaneous, neurological, psychiatric...), or a significant deviation from normal values observed during questioning, clinical examination or electrocardiogram (ECG);
* BMI > 30 (cardiovascular risk factor);
* Have a medical contraindication to sporting activities;
* Taking a medical treatment;
* Habitual sleep duration < 6 hours;
* Presenting a sleep disorder confirmed by questionnaire (Pittsburgh Sleep Quality Index Questionnaire > 5);
* Pregnant or breastfeeding
* Not covered by a health insurance plan;

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population is composed of healthy subjects .
Sampling Method: Non-Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Difference in average tracking accuracy on the simulator MATB-II depending on centrifuge acceleration (quantitative measurement) | Through study completion (26 months)
  MATB-II (Multi Attribute Task Battery) is a complex task simulator that mimics realistic tasks commonly performed by aircraft pilots during flight. Among these tasks, target tracking involves positioning a reticle at the center of the simulator's artificial horizon. The variance of the reticle's position as a function of the acceleration received in the centrifuge will be the primary outcome mesure in this study. This is a quantitative measure provided by the simulator.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de Recherche Biomédicale des Armées, Brétigny-sur-Orge, France

IPD SHARING:
Plan to Share IPD: Undecided